CLINICAL TRIAL: NCT02357537
Title: A Pilot Study Investigating a Decentralized Approach to Studying Dietary Intervention in Patients With Ulcerative Colitis
Brief Title: Decentralized Dietary UC Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Transparency Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TLS-UC-003
Record Dates: First submitted 2015-01-23; First posted 2015-02-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Colitis, Ulcerative
Keywords: Telemedicine
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional (Active Comparator): Subjects in Study Arm 1 will undergo a screening process, and if randomized, will follow a traditional, site-based clinical trial model and undergo a baseline visit and 3 more in-person visits with the Principal Investigator (total of 4 visits).
  Subjects in each Study Arm will be randomized (2:1) to follow one of two dietary regimens during the study: the Combined Anti-Inflammatory Diet (CAID) or Control (standard nutritional advice).
  Interventions: Behavioral: Combined Anti-inflammatory Diet (CAID)
- Remote (Active Comparator): Subjects in Study Arm 2 will undergo a screening process, and if randomized, will undergo one Baseline visit at the local Gastroenterologist's office and 4 video visits with the Principal Investigator. A mobile nurse will visit subjects at a distant location (such as their home) to obtain blood samples at visits 1 and 4.
  Subjects in each Study Arm will be randomized (2:1) to follow one of two dietary regimens during the study: the Combined Anti-Inflammatory Diet (CAID) or Control (standard nutritional advice).
  Interventions: Behavioral: Combined Anti-inflammatory Diet (CAID)

INTERVENTIONS:
Behavioral: Combined Anti-inflammatory Diet (CAID) — The CAID requires participants to modify their diet to include certain types of foods that may have anti-inflammatory properties. Participants on the CAID will be required to abstain from red meat and alcoholic beverages.

SUMMARY:
This study is designed to assess differences in remote and on-site patient study participation in the State of Massachusetts, as well as the significance of dietary interventions and their impact on UC. The study will activate one site with a Principal Investigator who will utilize each subject's local care system (local Gastroenterologist) to collect study data, along with telemonitoring and video visits, to make key study assessments and decisions regarding subjects' progression in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 and 80, inclusive, who reside in the state of Massachusetts.
2. Ability and willingness to provide documented informed consent and to comply with the study procedures, including in-person visits for Arm 1 and video visits for Arm 2.
3. Documented history of moderate to severe active UC
4. Disease duration of ≥12 weeks at the time of screening (diagnosed according to American College of Gastroenterology practice guidelines)
5. Screening fecal calprotectin>350 mg/g
6. Diagnosis of moderately to severely active UC, including historical endoscopy sub score ≥2; a rectal bleeding sub score ≥1 and disease activity a minimum of 25 cm from the anal verge.
7. Documented (via video or report) endoscopy performed within 2 years prior to randomization.
8. Access to a computer or mobile device with internet connection and an active email address.

Exclusion Criteria:

1. Prior extensive colonic resection, subtotal or total colectomy or planned surgery for UC
2. Past or present ileostomy or colostomy
3. Short bowel syndrome
4. Diagnosis of indeterminate colitis, fulminant colitis, toxic megacolon
5. Past or present fistula or abdominal abscess
6. History or current evidence of colonic mucosal dysplasia
7. Use of tube feeding, defined formula diets or parenteral alimentation/nutrition which has not been discontinued ≥3 weeks prior to study enrollment
8. Use of anticoagulants, herbal supplements and omega-3/fish oil supplements during the study
9. Crohn's Disease
10. Significant uncontrolled co-morbidity, such as neurological, cardiac (e.g., moderate to severe heart failure NYHA class III/IV), pulmonary, renal, hepatic, endocrine or gastrointestinal disorders
11. History of alcohol, drug or chemical abuse within 6 months prior to screening
12. Pregnant females, those intending to become pregnant, and those who are lactating
13. Current participation in any other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Endoscopy Mayo Score Comparison (proportion of endoscopies to which an independent reader can successfully assign an endoscopic Mayo Clinic sub-score) | Week 1
  Comparison of the proportion of endoscopies to which an independent reader can successfully assign an endoscopic Mayo Clinic sub-score between Study Arms 1 and 2.
Compliance (proportion of missing or non-evaluable records per patient and the proportion of patients who did not complete the study) | Week 7
  Comparison of the proportion of missing or non-evaluable records per patient and the proportion of patients who did not complete the study between Study Arms 1 and 2.
Combined Anti-inflammatory Diet (Change from baseline in fecal calprotectin/microbiome levels) | Weeks 0, 5 and 7
  Change from baseline in fecal calprotectin/microbiome levels between Control (standard nutritional advice) and CAID (dietary intervention) arms.

SECONDARY OUTCOMES:
Mayo Score and Patient Simple Clinical Colitis Activity Index Difference (Difference in partial Mayo Clinic sub-Score and Patient Simple Clinical Colitis Activity Index) | Weeks 1 and 7
  Difference in partial Mayo Clinic sub-Score and Patient Simple Clinical Colitis Activity Index between Control and CAID (dietary intervention).
Adverse Events | Weekly through week 11
  Difference in incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) between Study Arms 1 and 2 and between Control and CAID (dietary intervention) arms.
Dietary Compliance Comparison | Week 7
  Comparison of patient non-compliance events with dietary regimen between arms 1 and 2.
Participant Satisfaction Survey | Week 7
  Difference in reported patient satisfaction with trial participation between arms 1 and 2.
Mayo Score Discrepancy Frequency | Week 7
  Frequency of discrepancy between Principal Investigator-assessed and gastroenterologist-assessed Mayo Clinic Endoscopy Sub-Scores for Arm 2 patients at baseline.
Physician's Global Assessment Discrepancy Frequency | Week 7
  Frequency of discrepancy between Principal Investigator-assessed and gastroenterologist-assessed Mayo Clinic Physician's Global Assessment Sub-Score for Arm 2 patients at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Sablinski, MD, PhD, Study Director — Transparency Life Sciences
Locations (1):
- Crohn's and Colitis Center at Brigham and Women's Hospital, Brookline, Massachusetts, United States